CLINICAL TRIAL: NCT00775281
Title: Mediators of Neurogenic Inflammation in the Urinary Tract as Key Factors in the Painful Bladder Syndrome / Interstitial Cystitis and Bladder Dysfunction
Brief Title: Changes in Inflammatory and Contractile Protein Expression in Patients With Painful Bladder Syndrome/IC.
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: PD PhD K. Monastyrskaya, Institute of Anatomy, Balzerstrasse 2, 3000 Bern 9
Other Study IDs: KEK_146_05
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Overactive Bladder; Painful Bladder Syndrome; Chronic Pelvic Pain Syndrome; Cystitis, Interstitial
Keywords: Tachykinin receptors; Protein expression; Contractile proteins; Inflammatory proteins
MeSH Terms: conditions — Urinary Bladder, Overactive; Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — cold cut bladder biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1
- 2
- 3

SUMMARY:
Interstitial cystitis (IC)/chronic pelvic pain syndrome (CPPS) is a clinical syndrome of pelvic pain and/or urinary urgency/frequency in absence of a specific cause such as bacterial infection or damage to the bladder. The pathogenetic mechanisms of IC/CPPS are as yet undefined and it is largely this lack of knowledge, which precludes a systematic therapeutic approach. Experimental evidence, including results from the animal models of cystitis and the knock-out mice, indicate a participation of tachykinin receptors, especially the NK1R, in neurogenic inflammation, which is considered an important element of the IC complex. However, there is very scant information about the molecular mechanisms of IC in humans, or of the types of receptors, which participate in neurogenic inflammation. Based on our molecular biological know-how and the clinical expertise, we propose to investigate the role of the tachykinin and bradykinin receptors and their signalling partners in CPPS and bladder dysfunction in humans.

DETAILED DESCRIPTION:
Although IC has been recognised for more than a century, its pathophysiology remains a mystery, and as a consequence the treatment of IC is largely empirical. A multitude of mechanisms of the disease have been postulated ranging from neuroinflammatory to autoimmune or possibly infectious or toxic agents. Newer studies have hinted towards a genetic basis of the disease, but in most hypotheses an inflammatory component of some kind is involved and many findings support this theory. An often-cited hypothesis is the leaky epithelium. The healthy bladder is coated with a thin mucinous substance bladder surface mucin, which is composed of numerous sulfonated glycosaminoglycans and glycoproteins. In IC patients, in contrast to controls, as well as in some animal models of IC, qualitative changes to this surface layer have been observed (Lilly et al, 1990., Moskowitz et al, 1994). An initiating event (toxin) may lead to functional changes and increased permeability. This in turn leads to nerve sensitisation and possibly up-regulation. There is increasing evidence that the progression of IC is accompanied by a significant up-regulation of sensory nerves in the bladder (Letourneau, 1996). Nerve growth factor (NGF), a neurotropin that sensitises nociceptor fibres, was reported to be increased in bladders of IC patients (Lowe, 1997), and application of NGF in Wistar rats acutely induced bladder hyperactivity (Chuang, 2001). Sensory nerves in neurogenic inflammation secrete inflammatory mediators such as Substance P (SP), a nociceptive neurotransmitter in the central and peripheral nervous system. Increased amounts of the released Substance P have been found in the urine of IC patients (Hohenfellner, et al,1992, Pang et al., 1995, Pang et al., 1996), the concentration of Substance P reflecting the patients' degree of pain (Chen et al., 1999). Substance P and related tachykinins (TKs) mediate a variety of physiological processes in the genitourinary, pulmonary and gastrointestinal tract through stimulation of NK1 and NK2 receptors. Pre-clinical evidence obtained through use of selective tachykinin receptor antagonists indicates that endogenous tachykinins are involved in regulation of smooth muscle contraction, vasodilation, water metabolism and inflammation. Recently it was shown that mRNA encoding for SP receptor NK1 is in-creased in the bladder biopsies from patients with interstitial cystitis (Marchand et al., 1998). NK1R mRNA was found in detrusor muscle, urothelium and vascular structures, and the endothelial NK1R were markedly increased. SP binding to NK1R on endothelial cells results in vasodilation, plasma extravasation, cytokine release and activation and infiltration of immune cells, all characteristic of IC. Experiments with the NK1R knockout mice allowed for the first time to demonstrate the obligatory requirement of NK1R in cystitis and participation of these receptors in the chain of events linking mast cell degranulation and inflammation (Saban et al., 2000).

Changes in the sarcolemma, and altered expression of the tachykinin and bradykinin receptors might significantly influence the downstream signalling events leading to propagation of the symptoms of chronic pelvic pain/IC. By uncovering the link between clinical symptoms and the molecular regulation of the atypical inflammatory response, we may be able to offer novel and specific options for treatment. In the current proposal, we would like to further our studies of urinary bladder pathology, in particular the symptomatic complex of PBS/interstitial cystitis, and investigate the effect of changes in human urothelium and detrusor muscle cells on the NK1R-mediated signalling.

Biopsies from controls and PBS patients will be obtained in either general or spinal anesthesia transurethrally from the bladder dome and trigone with a biopsy tong. RNA will be extracted, and the expression levels of selected genes analyzed using Taqman real-time PCR and gene expression arrays (Applied Biosystems). Calcium imaging will be used to monitor the receptor activation and protein levels analysed by SDS-PAGE and Western Blotting. Receptor tissue distribution will be analysed by immuno-cytochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Clinical asymptomatic bladder function
* Clinical urgency frequency syndrome/ overactive bladder
* Clinical painful bladder syndrome/interstitial cystitis

Exclusion Criteria:

* Not able to understand patient information
* Other cause of symptoms
* Confusable diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: university hospital clinic
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Receptor expression in disease states versus control | at time of biospy

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Urology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Lilly JD, Parsons CL. Bladder surface glycosaminoglycans is a human epithelial permeability barrier. Surg Gynecol Obstet. 1990 Dec;171(6):493-6. PMID 2244283
- [Background] Letourneau R, Pang X, Sant GR, Theoharides TC. Intragranular activation of bladder mast cells and their association with nerve processes in interstitial cystitis. Br J Urol. 1996 Jan;77(1):41-54. doi: 10.1046/j.1464-410x.1996.08178.x. PMID 8653316
- [Background] Lowe EM, Anand P, Terenghi G, Williams-Chestnut RE, Sinicropi DV, Osborne JL. Increased nerve growth factor levels in the urinary bladder of women with idiopathic sensory urgency and interstitial cystitis. Br J Urol. 1997 Apr;79(4):572-7. doi: 10.1046/j.1464-410x.1997.00097.x. PMID 9126085
- [Background] Chuang YC, Fraser MO, Yu Y, Chancellor MB, de Groat WC, Yoshimura N. The role of bladder afferent pathways in bladder hyperactivity induced by the intravesical administration of nerve growth factor. J Urol. 2001 Mar;165(3):975-9. PMID 11176525
- [Background] Hohenfellner M, Nunes L, Schmidt RA, Lampel A, Thuroff JW, Tanagho EA. Interstitial cystitis: increased sympathetic innervation and related neuropeptide synthesis. J Urol. 1992 Mar;147(3):587-91. doi: 10.1016/s0022-5347(17)37314-7. PMID 1538434
- [Background] Pang X, Marchand J, Sant GR, Kream RM, Theoharides TC. Increased number of substance P positive nerve fibres in interstitial cystitis. Br J Urol. 1995 Jun;75(6):744-50. doi: 10.1111/j.1464-410x.1995.tb07384.x. PMID 7542136
- [Background] Pang X, Boucher W, Triadafilopoulos G, Sant GR, Theoharides TC. Mast cell and substance P-positive nerve involvement in a patient with both irritable bowel syndrome and interstitial cystitis. Urology. 1996 Mar;47(3):436-8. doi: 10.1016/S0090-4295(99)80469-5. PMID 8633418
- [Background] Marchand JE, Sant GR, Kream RM. Increased expression of substance P receptor-encoding mRNA in bladder biopsies from patients with interstitial cystitis. Br J Urol. 1998 Feb;81(2):224-8. doi: 10.1046/j.1464-410x.1998.00507.x. PMID 9488063
- [Background] Moskowitz MO, Byrne DS, Callahan HJ, Parsons CL, Valderrama E, Moldwin RM. Decreased expression of a glycoprotein component of bladder surface mucin (GP1) in interstitial cystitis. J Urol. 1994 Feb;151(2):343-5. doi: 10.1016/s0022-5347(17)34944-3. PMID 8283520
- [Background] Saban R, Saban MR, Nguyen NB, Lu B, Gerard C, Gerard NP, Hammond TG. Neurokinin-1 (NK-1) receptor is required in antigen-induced cystitis. Am J Pathol. 2000 Mar;156(3):775-80. doi: 10.1016/S0002-9440(10)64944-9. PMID 10702392